CLINICAL TRIAL: NCT07379502
Title: Endometrial Response in Women With Poorly Primed Endometrial Lining in Diagnosed Polycystic Ovarian Syndrome Treated With Letrozole Alone or With Added Estradiol Valerate
Brief Title: Endometrial Response in Polycystic Ovarian Syndrome Treated With Letrozole Alone or With Added Estradiol Valerate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Kharian Medical College (Other Government)
Responsible Party: Principal Investigator, Maryum Noor Malik, Senior Registrar Ob/Gyn, CMH Kharian Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKMC/IERB/AC-00256
Record Dates: First submitted 2025-11-26; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: PCOS (Polycystic Ovary Syndrome); Letrozole; Estradiol Valerate; Endometrial response; Endometrial thickness
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Aromatase Inhibitors; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- letrozole (Active Comparator): 30 participants with PCOs will receive tab letrozole 2.5mg 2 x OD for 5 days
  Interventions: Drug: Letrozole (Aromatase Inhibitors)
- letrozole plus estradiol valerate (Experimental): 30 participants with PCOs will receive tab letrozole 2.5mg 2 x OD for 5 days plus tab Estradiol valerate 2mg OD for 12 days
  Interventions: Drug: Letrozole (Aromatase Inhibitors) + Estradiol valerate

INTERVENTIONS:
Drug: Letrozole (Aromatase Inhibitors) — 30 participants with PCOs will receive tab letrozole 2.5mg 2 x OD for 5 days
  Arms: letrozole
Drug: Letrozole (Aromatase Inhibitors) + Estradiol valerate — 30 participants with PCOs will receive tab letrozole 2.5mg 2 x OD for 5 days plus tab Estradiol valerate 2mg OD for 12 days
  Arms: letrozole plus estradiol valerate

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is one of the most common endocrine disorders among women of reproductive age, characterized by chronic anovulation, hyperandrogenism, and polycystic ovarian morphology. Letrozole, an aromatase inhibitor, has emerged as a first-line ovulation induction agent due to its superior ovulation and pregnancy rates compared to clomiphene citrate. Estradiol valerate, a synthetic estrogen, can be co-administered with letrozole to improve endometrial receptivity by enhancing endometrial thickness, vascularity, and pattern. This study aims to evaluate the effect of letrozole alone versus letrozole with estradiol valerate on endometrial development in these patients.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is one of the most common endocrine disorders among women of reproductive age, characterized by chronic anovulation, hyperandrogenism, and polycystic ovarian morphology. Letrozole, an aromatase inhibitor, has emerged as a first-line ovulation induction agent due to its superior ovulation and pregnancy rates compared to clomiphene citrate. However, one of the drawbacks of aromatase inhibitors is suboptimal endometrial development, which may adversely affect implantation and pregnancy outcomes.

Estradiol valerate, a synthetic estrogen, can be co-administered with letrozole to improve endometrial receptivity by enhancing endometrial thickness, vascularity, and pattern. Limited data exist on whether adding estradiol to letrozole truly improves the endometrial response and clinical pregnancy rates in women with PCOS. This study aims to evaluate the effect of letrozole alone versus letrozole with estradiol valerate on endometrial development in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-35 years
* Clinical diagnosis of PCOS (Rotterdam criteria)

Exclusion Criteria:

* Endocrine disorders other than PCOS
* Endometrial pathology or uterine malformations
* Allergy to letrozole or estradiol
* Hormonal therapy within last 3 months

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness (mm) on day of ovulation trigger | 12th day of cycle 1 (Each cycle is 28 days)
  Endometrial thickness will be measured on Transvaginal ultrasound on 12th day in a 28 day menstrual cycle.
Pattern of endometrium (Trilaminar or Non-trilaminar) on the day of ovulation trigger | 12th day of cycle 1 (Each cycle is 28 days)
  Endometrial pattern will be seen on Transvaginal ultrasound on 12th day in a 28 day menstrual cycle

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Kharian Medical College, Khārian, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No